CLINICAL TRIAL: NCT06304714
Title: Abnormalities of Plasma Willebrand Factor Activity Induced by Bothrops Snakebites Endemic to Martinique and French Guyana
Brief Title: Effects of Bothrops Spp. Snake Envenomation on Willebrand Factor Activity in Martinique and French Guiana
Acronym: WBOTHROPS
Status: Recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 20_RIPH3-16; 2022-A00162-41 (Other: ANSM (National Agency for the Safety of Medicines and other health products ))
Record Dates: First submitted 2024-02-19; First posted 2024-03-12 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Snake Envenomation; Thrombi; Coagulopathy; Hemorrhage
Keywords: Snakebite envenomation; French Caribbean (Martinique, French Guiana); Bothrops species; Von Willebrand Factor; endothelial activity; haemostasis
MeSH Terms: conditions — Snake Bites; Thrombosis; Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A plasma library will be set up during this research with the aim of carrying out subsequent analyses (research projects on Bothrops bites in Martinique and French Guiana, with planned collaborations on a regional and international scale).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient from french Guiana: 15 patients suffering from envenomation by Bothrops bites endemic to French Guiana
  Interventions: Other: Patients suffering from envenomation by Bothrops
- Patient from Martinique: 15 patients suffering from envenomation by Bothrops Lanceolatus bites endemic to Martinique.
  Interventions: Other: Patients suffering from envenomation by Bothrops

INTERVENTIONS:
Other: Patients suffering from envenomation by Bothrops — For research purposes, the investigator will collect six additional tubes of blood during a venipuncture. This additional volume of blood will be used for research analysis.
  The total volume drawn will be within the maximum volume of blood that can be drawn based on body weight.
  Venous sampling is planned as part of routine care and the additional blood volumes collected are not significant. This is a low risk procedure due to the small amount of extra blood taken (25,5 ml).

SUMMARY:
In 2017, the World Health Organization placed snakebites at the top of its list of neglected tropical diseases in an effort to facilitate funding for prevention programs, improve access to anti-venom, and stimulate new research in this area. Between 5 and 25 cases per 100 000 inhabitants are reported per year in French Guiana and Martinique. Before the era of anti-venom immunotherapy, envenomations by Bothrops snake bites in French Guiana and Martinique could quickly become life-threatening with a mortality rate close to 30%. Today, the administration of fragments of Fab or (Fab')2 immunoglobulins gives anti-venoms an excellent capacity to neutralise venom toxins, which has reduced mortality to less than 1% in the case of early hospital treatment In French Guiana, envenomation by Bothrops bites is characterized by local signs such as intense pain, rapidly expanding oedema, haemorrhagic phlyctenes and sometimes muscle necrosis. The local inflammatory and haemorrhagic damage is related to the enzymatic activities of the toxins contained in the venom (metallo-proteinases, disintegrins, and phospholipases A2, in particular). At the systemic level, venom serine proteases and metalloproteinases activate the coagulation cascade by multiple mechanisms (activation of coagulation factors X and V and of protrombin, thrombin-like and fibrinogenolytic enzymatic properties) and are responsible for the collapse of coagulation factors making the blood incoagulable. The metalloproteinases "hemorrhagins" destroy the vessel wall and are the cause of locoregional and systemic hemorrhage.

Envenomations by bites of Bothrops lanceolatus in Martinique have particular characteristics. Despite the genetic similarity with their congeners in French Guiana, envenomation by bites of Bothrops lanceolatus is characterized by the development of very intense local inflammatory signs (little haemorrhage) and the occurrence of thrombotic complications such as cerebral, pulmonary or myocardial infarction. The mechanisms behind this thrombotic presentation are not known. The large amount of metalloproteinases in the composition of Bothrops lanceolatus venom is believed to be responsible for destruction of vascular endothelium and pro-thrombotic state. Bothrops lanceolatus bite envenomations have been reported to be frequently complicated by generalized infections, disseminated intravascular coagulation and the occurrence of multi-visceral failure syndrome. This observation suggests abnormalities in endothelial function in which changes in Willebrand factor expression have been implicated.

The investigators hypothesize that plasma Willebrand factor (VW) activity and the intensity of endothelial activation are different depending on the Bothrops snake species involved in the bites in Guyana and Martinique. Due to the specific properties of the venoms of each Bothrops species, the activity of the Willebrand factor (VW) and the consequences in terms of endothelial activation would be different and responsible for the clinico-biological characteristics according to the geographical origin of the snakes.

The investigators will demonstrate that the accumulation of Willebrand factor (VW) and the increase in its activity are responsible for the endothelial activation and micro-thrombosis observed during envenomations by Bothrops lanceolatus bites, whereas the decrease in its activity induced by the venoms of endemic Bothrops from Guyana is responsible for haemorrhagic phenomena.

This study will highlight the importance of changes in Willebrand factor activity on endothelial activation and the initiation of micro-thrombosis in the case of Bothrops lanceolatus envenomations and on primary haemostasis and bleeding disorders in the case of endemic Bothrops in Guyana. This new knowledge is important insofar as individualised therapeutic management can be proposed. Indeed, several studies have shown that adjuvant treatment of thrombotic microangiopathies, such as thrombotic thrombocytopenic purpura, with blood products (fresh frozen plasma) or plasma exchange, improves endothelial dysfunction and the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women, at least 18 years old
* Be admitted to the Emergency Department of the Martinique University Hospital or the Cayenne University Hospital
* Be the victim of a confirmed Bothrops snake bite in Martinique or French Guyana. The formal identification of the snake by the patient or his entourage is imperative.
* Have a confirmed diagnosis of stage III envenomation (regional oedema of the limb and/or moderate general symptoms such as moderate hypotension, malaise, vomiting, abdominal pain, diarrhoea) and stage IV (extensive oedema reaching the trunk and/or severe general symptoms such as prolonged hypotension, shock, anaphylactoid reaction, visceral damage)
* Be able to receive and understand information related to the research
* Be able to freely give verbal consent to participate in the proposed research
* Be able to freely give written informed consent to participate in the plasmathèque
* Be affiliated to the general social security system

Exclusion Criteria:

* Pregnant or breastfeeding woman
* People who have been treated for snakebite with Bothrops anti-venom Bothrofav® or Antivipmyn-tri®.
* Known disorders of haemostasis such as haemophilia A (factor VIII deficiency), haemophilia B (factor IX deficiency), vitamin K deficiency, hepato-cellular insufficiency, presence of circulating anticoagulant factors
* Disseminated intravascular coagulation (DIC)
* Constitutional and acquired Von Willebrand disease
* Constitutional and acquired thrombopathies
* Idiopathic thrombocytopenic purpura
* Person under legal protection (guardianship, curatorship, safeguard of justice), and person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients hospitalized in the emergency and intensive care units of the Martinique University Hospital or the Cayenne University Hospital (French Guiana).
  Patient recruitment will be organized by center throughout the 18-month study period.
  Initial data collection (D0) will be carried out on admission to the hospital ward, using a blood sample taken as part of the treatment and for research purposes, to collect indicators relating to plasma Willebrand factor activity and the endothelial response induced by Bothrops bites. These indicators collected on D0 will constitute the reference data specific to each individual. At D1 and D8, these indicators will be collected again.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Plasma Willebrand factor (VW:Act) activity prior to administration of the anti-venom (Bothrofav® or Antivipmyn-tri®). | Day 0 (initail hospital admission)
  VW:Act will be compared according to the type of Bothrops species involved (Martinique vs French Guiana)

SECONDARY OUTCOMES:
Plasma VW factor activity (VW:Act/VW:Ag ratio) | Day 1 and day 8
  VW activity (VW:Act) will be standardized according to its antigenic expression (VW:Ag). Hence, the outcome measure 2 will be the ratio VW:Act/VW:Ag.
  This outcome measure will be compared according to the endemic origin of the Bothrops species (Martinique or French Guiana).

OTHER OUTCOMES:
Hemostasis abnormalities | Day 0, day 1 and day 8
  Hemostasis abnormalities measured will be:
  * blood count and platelet count
  * thrombin time (PT)
  * activated partial thromboplastin time (APTT)
  * fibrinogen level
  * fibrin monomer and fibrin degradation product (D-dimer) levels These different hemostasis abnormalities will be compared according to the endemic origin of the Bothrops species (Martinique or French Guiana).
Plasma levels of high-molecular-weight VW factor multimers assessed by electrophoresis technique | Day 0, day 1 and day 8
  This outcome measure will be compared according to the endemic origin of the Bothrops species (Martinique or French Guiana).
Plasma concentrations of soluble forms of the endothelial adhesion molecules | Day 0, day 1 and day 8
  The plasma concentrations (measured by ELISA technique) of the following endothelial adhesion molecules will be analyzed:
  * ICAM-1,
  * VCAM-1
  * E-selectins All endothelial adhesion molecule concentrations will be compared according to the endemic origin of the Bothrops species (Martinique or French Guiana).

CONTACTS AND LOCATIONS:
Overall Officials: REMI NEVIERE, Professor, Study Director — University Hospital of Martinique; DABOR RESIERE, Professor, Principal Investigator — University Hospital of Martinique; HATEM KALLEL, Professor, Principal Investigator — Hospital of Cayenne, FRENCH GUIANA
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, Martinique, Martinique

IPD SHARING:
Plan to Share IPD: No